CLINICAL TRIAL: NCT05363527
Title: Experimental Model of Depression in Aging: Anxiety, Inflammation, and Reward Mechanisms
Brief Title: Aging and Reward System Response to Inflammation and Anxiety Study
Acronym: ARIA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Chloe Boyle, PhD, Adjunct Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: K01AG072049 (NIH); 1K01AG072049-01A1 (NIH)
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Anhedonia; Inflammation; Anxiety; Aging; Depression
Keywords: anxiety; aging; anhedonia; inflammation
MeSH Terms: conditions — Anhedonia; Inflammation; Anxiety Disorders; Depression | interventions — Endotoxins

STUDY DESIGN:
Intervention Model Description: Endotoxin vs. Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Endotoxin (Experimental): Endotoxin 0.8 ng/kg body weight
  Interventions: Biological: Endotoxin
- Placebo (Placebo Comparator): same volume of 0.9% saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Endotoxin — Endotoxin
  Arms: Endotoxin
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to use an experimental inflammatory challenge to examine whether older adults with symptoms of anxiety experience loss of pleasure or loss of motivation when they are exposed to inflammation. Loss of pleasure or loss of motivation will be evaluated using self-report questionnaires, computer tasks, and during a brain scan.

DETAILED DESCRIPTION:
Participants will undergo phone screening, two in-person visits, and telephone follow-up. The first visit will last 4 hours and the second visit will last 10.5 hours. Phone screening and follow-up will take no longer than 30 minutes.

Phone Screening and Visit #1:

Following phone screening to determine potential eligibility, participants will have an in-person evaluation. Following informed consent in the first session, participants will undergo semi-structured clinical interviews and complete questionnaires to assess medical- and medication histories; current- and past history of psychiatric disorders, and evaluation of behavioral symptoms of anxiety and depression. They will also complete computer tasks that assess motivation and sensitivity to reward. As part of one of these tasks, they will be asked to provide a picture of a loved one, which they will later view during a fMRI scan.

Visit #2 and telephone follow-up:

The second session will be about two weeks later. It will begin at 7:30AM and will involve placement of two intravenous catheters (one in each arm), evaluation of heart rate and blood pressure, administration of endotoxin vs. placebo, repeated blood sampling along with questionnaires about mood and symptoms for approximately 10.5 hours. Two hours post-injection participants will complete a 1-hour brain scan that includes tasks to assess motivation and sensitivity to reward. Study staff will escort the participant to a nearby facility to complete the brain scan. 24 hrs and 2-weeks following this session, study staff will call the subject and ask about physical and mood symptoms, using the same set of items used during the experimental protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be required to be in good general health (as evaluated during the phone and in-person baseline session)
* Participants will be aged 60 to 80 years.
* 3/4 the participants (n=30) will be those with clinically significant anxiety as defined by a score of 5 or greater on the GAD-7;
* 1/4 the participants (n=10) will be those with low anxiety as defined by a GAD-7 score of <5.

Exclusion Criteria:

* Presence of chronic mental or physical illness (except for anxiety)
* History of allergies, autoimmune, liver, or other severe chronic diseases
* Current and regular use of prescription medications such as steroids, non-steroid anti-inflammatory drugs, aspirin, immune modifying drugs, opioid analgesics, statins, antihypertensive drugs, anti-arrhythmic drugs, and antidepressant medications (none in the last 6 months)
* Nightshift work or time zone shifts (> 3hrs) within the previous 6 weeks
* Previous history of fainting during blood draws.
* Claustrophobia
* Metal in the body
* Presence of co-morbid medical conditions not limited to but including cardiovascular (e.g., history of acute coronary event, stroke) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders;
* Presence of comorbid inflammatory disorders such as rheumatoid arthritis or other autoimmune disorders;
* Presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or to put the study participant at undue risk;
* Presence of chronic infection, which may elevate pro-inflammatory cytokines;
* Presence of an acute infectious illness in the two weeks prior to an experimental session.
* Current Axis I psychiatric disorders other than anxiety as determined by the Research Version of the Structured Clinical Interview
* Lifetime history of suicide attempt or inpatient psychiatric admission.
* Sleep Disorders: Current history of sleep apnea or nocturnal myoclonus;
* Phase-shift disorder
* Current and/or past regular use of hormone-containing medications including steroids;
* Current and/or past regular use of non-steroid anti-inflammatory drugs;
* Current and/or past regular use of immune modifying drugs that target specific immune responses such as cytokine antagonists;
* Current and/or past regular use of analgesics such as opioids;
* Current and/or past regular use of cardiovascular medications, including antihypertensive, anti-arrhythmic, antianginal, and anticoagulant drugs;
* Current smoking
* Current excessive caffeine use (>600 mg/day) because of the known effects on pro-inflammatory cytokine levels;
* Evidence of recreational drug use from urine test.
* Body mass index > 35 because of the effects of obesity on proinflammatory cytokine activity
* Any clinically significant abnormality on screening laboratory tests
* Clinically significant abnormalities in electrocardiogram

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Neural Indices of Reward Motivation - Anticipatory Reward Response | approximately 2 hours post-injection for 7 minutes
  Task-based functional magnetic resonance imaging (fMRI) will be used to assess reward motivation, as operationalized by ventral striatum (VS) activity during anticipation of monetary reward cue trials vs no-reward cue trials during the Monetary Incentive Delay Task.
Neural Indices of Reward Motivation - Effort-Based Decision Making | approximately 2 hours post-injection for 14 minutes
  Task-based functional magnetic resonance imaging (fMRI) will be used to assess effort-based motivational processing, as assessed by VS, ventromedial prefrontal cortex (vmPFC), and pre-supplementary motor area (pre-SMA) activity with choice phase as event onset during an adapted version of the Effort Expenditure for Rewards Task (EEfRT).
Neural Indices of Monetary Reward Sensitivity during Effort-Based Decision Making | approximately 2 hours post-injection for 14 minutes
  Task-based functional magnetic resonance imaging (fMRI) will be used to assess sensitivity for monetary reward, as operationalized by VS and VMPFC activity during receipt of monetary reward (vs. fixation) and during choice of low vs. high reward trials during the EEfRT.
Neural Indices of Reward Sensitivity for Non-Monetary Reward | approximately 2 hours post-injection for 10 minutes
  Sensitivity for non-monetary reward as assessed by VS and VMPFC activity when viewing positive non-social vs neutral images, and when viewing positive social vs. neutral images, in a positive picture viewing task.

SECONDARY OUTCOMES:
Resting state functional connectivity | 2 hours post-injection for 7 minutes
  Resting-state functional connectivity will be assessed over a 7-minute period, focusing on functional connectivity between the ventromedial prefrontal cortex and ventral striatum.
Social Incentive Delay Task - Neural Indices of Social Reward Motivation | approximately 2 hours post-injection for 7 minutes
  Task-based functional magnetic resonance imaging (fMRI) will be used to assess social reward motivation, as operationalized by ventral striatum (VS) activity during anticipation of social reward cue trials vs no-reward cue trials on the Social Incentive Delay Task.
Social Incentive Delay Task - Neural Indices of Reward Motivation for Close Social Reward | approximately 2 hours post-injection for 7 minutes
  Motivational processing for a close other social reward will be assessed with the Social Incentive Delay Task as VS activity during anticipation of viewing images of a close other (vs no-reward cue).
Behavioral Indices of Reward motivation - close other social reward | 2 hours post-injection
  Motivational processing for a close other social reward will be assessed as self-reported desire to be around the close other on a scale of 1 (not at all) to 7 (a lot).
Monetary Incentive Delay Task -Neural Indices of Monetary Reward Sensitivity | approximately 2 hours post-injection for 7 minutes
  Sensitivity for monetary reward as assessed by VS and VMPFC activity during outcome (reward vs. no-reward) and anticipation (low vs. high reward cues) on the Monetary Incentive Delay task.
Social Incentive Delay Task - Neural Indices of Social Reward Sensitivity | approximately 2 hours post-injection for 7 minutes
  Sensitivity for social reward as assessed by VS and VMPFC activity during outcomes (reward vs. no-reward) on the Social Incentive Delay Task.
Social Incentive Delay Task - Neural Indices of Reward Sensitivity for Close Social Reward | approximately 2 hours post-injection for 7 minutes
  Reward sensitivity for a close other will be assessed as VS and VMPFC activity during the outcome phase (close other reward vs no-reward outcomes) and anticipation phase (general social reward vs. close other social reward cue anticipation) on the Social Incentive Delay Task.
Behavioral Indices of Reward Motivation - Effort-Based Decision Making | Pre-injection and approximately 2 hours post-injection
  Motivation for monetary reward is assessed with an Effort Expenditure for Rewards Task (EEfRT); willingness to exert physical effort for monetary reward (i.e., selection of hard vs easy tasks) is the outcome measure with higher willingness indicative of higher motivation.
Behavioral Indices of Reward Sensitivity and Learning - Probabilistic Reward Task | Pre-injection and approximately 2 hours post-injection
  Implicit reward learning and sensitivity to monetary reward is assessed with the probabilistic reward task (PRT); change in the magnitude of response bias from baseline to post-injection is the outcome measure. Higher response bias indicates higher reward sensitivity/learning.
Depressed Mood Subscale of the Profile of Mood States (POMS) | 10 hours
  The Depressed Mood Subscale of the POMS is a self-reported assessment of depressed mood in which subjects rate severity of depressed mood using a visual analog scale from 1 to 10 (10 being most severe). Each timepoint is scored and analyses examine the temporal profile of change with assessment every hour
Motivation for social and non-social reward (interest in activities scale). | 10 hours
  This task will evaluate motivation for reward by subjective reports of interest in engaging in a variety of social and non-social activities on a 1 to 5 Likert scale on an hourly basis, with higher score indicating more interest. Each timepoint is scored and analyses examine the temporal profile of change with assessment at baseline and at 1 hour intervals post-injection.

OTHER OUTCOMES:
Behavioral Indices of Reward Motivation and Sensitivity with Incentive Delay Tasks | approximately 2 hours post-injection for 14 minutes
  Behavioral performance on the Monetary and Social Incentive Delay Tasks is tested as reaction time for reward vs no- reward cue trials (an index of motivation) and reaction time for low vs. high reward trials (an index of sensitivity to changes in reward magnitude).
Behavioral Indices of Reward Sensitivity - Positive Images Task | approximately 2 hours post-injection for 10 minutes
  Sensitivity for non-monetary reward assessed by self-report affect when viewing positive non-social vs neutral images, and when viewing positive social vs. neutral images, on a 1(extremely negative affect) to 4(extremely positive affect) scale.
Behavioral Indices of Reward Sensitivity - EEfRT | Pre-injection and 2 hours post-injection
  Sensitivity for monetary reward assessed by the degree to which higher potential winnings predict hard task choice.
Emotion Intensity Task | Baseline and 3 hours post-injection for five minutes
  This is a short computer-based task used to test emotion detection with a face morphing task. Faces morph from neutral to expressions of emotions (happy, sad, angry, or fearful) and participants indicate when and what emotion is presented; the dependent variables are reaction time and accuracy.
Attentional Bias Task | Baseline and 3 hours post-injection for five minutes
  This is a short computer-based task used to test attentional bias towards positive and negative valenced facial expressions (low arousal happy, high arousal happy, sad, angry) relative to neutral faces. Higher attentional bias scores indicate greater bias towards emotion.
Systemic marker of inflammation as indexed by interleukin-6. | 10 hours
  Systemic inflammation as measured by circulating levels of interleukin-6 in plasma in pg/ml. Each timepoint is assayed and analyses examine the temporal profile of change with assessment every hour
Genomic marker of inflammation | baseline and .5, 1, and 2 hours post-injection
  Transcriptional profile of inflammation as measured by Conserved Translational Response to Adversity in circulating peripheral blood mononuclear cells
Executive function - inhibition with the antisaccade task. | Baseline and 4 hours post-injection for 10 minutes.
  The Antisaccade task is used to assess Inhibition. Participants are tasked with inhibiting a reflexive response towards a visual cue in order to correctly identify a target stimulus presented elsewhere. For each of 72 trials, participants view a centrally positioned fixation point (the letter X) on the computer screen for a variable amount of time (1500-3500ms). A visual cue (a black circle) is then presented on one side of the computer screen for 225ms. The target stimulus (a number from 1 to 9) is presented on the opposite side of the screen for 250, 233, or 200ms before being masked by gray cross-hatching. The participant verbally reports the target number to a trained research assistant or recording device or uses the keyboard to indicate the number. The participant does not receive feedback regarding accuracy, and there is no time limit for participant response for each trial.
Executive function - updating with the spatial 2-back task | Baseline and 4 hours post-injection for 10 minutes.
  The Spatial 2-Back task is used to assess Updating, the ability to monitor and replace information in working memory. For each of 120 trials, participants view an array of boxes, 11 white and 1 black. The location of the black box varies across trials. Participants are tasked with using one of two keys to indicate whether the black box is presented in the same location as it was two trials back. Participants do not receive feedback regarding accuracy, and trials proceed automatically if a response is not made within 2000ms. The task includes 20 practice trials
Executive function - shifting with color-shape task. | Baseline and 4 hours post-injection for 10 minutes.
  The Color-Shape task is used to assess Shifting, or the ability to switch between mental sets. For each of 104 trials, participants are presented with a circle or square that is of blue or red color. Participants are asked to use 1 of 2 keys to indicate whether the figure is red or blue (52 color trials) or square or triangle (52 shape trials). One key is paired with a color and a shape (e.g., red and square) and one key is paired with the other color and shape (e.g., blue and circle). For each trial, the letter C or S is presented above the figure to indicate color versus shape trials. The order of C/S trials is randomized, and there is no time limit for participant response for each trial. A quiet "ding" occurs following incorrect trials. The task includes 52 practice trials: 26 color followed by 26 shape trials.
Depressed mood and depressive symptoms as measured by the Montgomery Asberg Depression Rating Scale (MADRS) | 10 hours
  Depressed mood and depressive symptom severity by self-reported assessment using the Montgomery Asberg Depression Rating scale with a range from 0 to 54 with a higher score indicating more severe depressive symptoms. Each timepoint is scored and analyses examine the temporal profile of change with assessment at baseline and at 2 hour intervals post-injection.

CONTACTS AND LOCATIONS:
Overall Officials: Chloe C Boyle, PHD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Norman Cousins Center for Psychoneuroimmunology, University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available to users upon request, provided the investigators are working under an institution with a Federal Wide Assurance (FWA). All requests for transfer of materials for research purposes will be made through a UCLA onlineMTA. Persons requesting access will be required to complete a data-sharing agreement providing for the maintenance of the confidentiality of research participants, describing use to which the data will be put, and requiring acknowledgement of the source of the data and its underlying NIA funding. The names and institutions of persons either given or denied access to the data, and the bases for such decisions, will be summarized in annual progress reports.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available by the on-line publication date once the data has been accepted for publication. All submitted data will conform to relevant data and terminology standards. This data sharing policy is intended to allow investigators sufficient time for data verification, and for submission of primary publications based on the collected data. We will identify where the data will be available, and how to access the data (i.e., by contacting Dr. Boyle directly), in any publication or presentation by Dr. Boyle and her mentorship team. Finally, we will acknowledge the funding source in any and all publications and presentations using these data.
Access Criteria: * investigators must be working under an institution with a Federal Wide Assurance (FWA);
  * persons requesting access will be required to complete a data-sharing agreement providing for the maintenance of the confidentiality of research participants, describing use to which the data will be put, and requiring acknowledgement of the source of the data and its underlying NIA funding.